CLINICAL TRIAL: NCT00589225
Title: Correlation of Disease Expression With Specific Genetic Mutations in Primary Hyperoxaluria
Brief Title: Primary Hyperoxaluria Mutation Genotyping
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Oxalosis and Hyperoxaluria Foundation (OHF) (Other)
Responsible Party: Principal Investigator, Dawn S. Milliner, M.D., M.D., Mayo Clinic
Other Study IDs: 434-03; R01DK073354 (NIH)
Record Dates: First submitted 2007-12-28; First posted 2008-01-09 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Primary Hyperoxaluria
Keywords: PH; PH type I; Primary Hyperoxaluria; Hyperoxaluria; Primary Oxalosis; PH type II; PH type III; Genetic testing for PH; Genetic testing for Primary Hyperoxaluria; Hereditary study for PH; Hereditary study for Primary Hyperoxaluria
MeSH Terms: conditions — Hyperoxaluria, Primary; Hyperoxaluria | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Genetic Analysis
  Interventions: Genetic: Genetic Analysis

INTERVENTIONS:
Genetic: Genetic Analysis — We will draw one tube of blood from your arm to obtain white blood cells. These white blood cells will be used as a source of DNA for genetic testing.

SUMMARY:
This study will help us determine whether certain genetic mutations, more than others, are a cause of more severe disease in Primary Hyperoxaluria.

DETAILED DESCRIPTION:
During your study visit, we will draw one tube, about two teaspoonfuls (1 to 1 ½ teaspoons for children), of blood from your arm to obtain white blood cells. These white blood cells will be used as a source of DNA for genetic testing. We will use the isolated DNA to try to identify the gene that is defective in Primary Hyperoxaluria by comparing it with the structure of genes in normal individuals, patients with Primary Hyperoxaluria, and family members of Primary Hyperoxaluria patients. In family members of primary hyperoxaluria patients, a 24 hour urine test may also be collected.

ELIGIBILITY:
Inclusion Criteria:

* You have been diagnosed, or you are in the process of being diagnosed Primary Hyperoxaluria
* You have a family member diagnosed with Primary Hyperoxaluria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with clinical findings suggestive of primary hyperoxaluria
  * Family members of patiente with clinical findings suggestive of primary hyperoxaluria
Sampling Method: Non-Probability Sample
Enrollment: 902 (Actual)
Dates: Start 2003-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To determine whether certain genetic mutations, more than others, are a cause of more severe disease in Primary Hyperoxaluria | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Milliner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Hyperoxaluria Center — http://www.mayoclinic.org/nephrology-rst/hyperoxaluriacenter.html
- See also: Mayo Clinic Hyperoxaluria and Oxalosis — http://www.mayoclinic.org/hyperoxaluria/